CLINICAL TRIAL: NCT04653623
Title: Effect of Tranexamic Acid on Blood Loss After High Tibial Osteotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Tranexamic Acid
Record Dates: First submitted 2020-10-20; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid before high tibial osteotomy (Experimental): Interventions
  * Procedure/Surgery: High tibial osteotomy
  * Drugs: Tranexamic acid
  Interventions: Procedure: High tibial osteotomy; Drug: Tranexamic acid
- High tibial osteotomy only (Active Comparator): Interventions
  - Procedure/Surgery: High tibial osteotomy
  Interventions: Procedure: High tibial osteotomy

INTERVENTIONS:
Procedure: High tibial osteotomy — Treatment option for medial compartment osteoarthritis of knee
Drug: Tranexamic acid — Medication used to treat or prevent excessive blood loss from major trauma, postpartum bleeding, surgery, tooth removal, nosebleeds, and heavy menstruation
  Arms: Tranexamic acid before high tibial osteotomy

SUMMARY:
This study aims to examine whether tranexamic acid has an meaningful clinical effect on blood loss after high tibial osteotomy. This study design is a double-blind randomized controlled trial. The patients were randomly assigned to intervention or usual care groups. Intervention patients receive tranexamic acid 2g for 10 minutes just before surgery. Primary outcome is hemoglobin level preoperatively, postoperative 1 day, 2 days, 3 days, 2 weeks. Secondary outcome included hematocrit level, hemovac drainage, total blood loss, need for transfusion, deep vein thrombosis, Visual Analog Pain Scale, and wound complication.

DETAILED DESCRIPTION:
High tibial osteotomy is proved treatment option for medial compartment osteoarthritis of knee joint. Especially, open wedge high tibial osteotomy might cause moderate amount of bleeding and hematoma formation. Bleeding and hematoma could be a reason of soft tissue infection and wound complications. Tranexamic acid (TXA) is a medication used to treat or prevent excessive blood loss from major trauma, postpartum bleeding, surgery, tooth removal, nosebleeds, and heavy menstruation. The objective of the study is to test whether preoperative tranexamic acid could reduce the postoperative complications due to bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Patients for high tibial osteotomy
* Having medicare insurance
* Accepted patients

Exclusion Criteria:

* History of lower extremity infection or neurologic problems
* Inflammatory arthritis
* Using thrombins
* History of treatment for anemia
* History of thromboembolic event
* Chronic kidney disease

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin level | Change from Baseline Hemoglbin level at postoperative 1 day
Hemoglobin level | Change from Baseline Hemoglbin level at postoperative 2 days
Hemoglobin level | Change from Baseline Hemoglbin level at postoperative 3 days
Hemoglobin level | Change from Baseline Hemoglbin level at postoperative 2 weeks

SECONDARY OUTCOMES:
Hematocrit level | Preoperative & postoperative 1, 2, 3 days, 2 weeks
Amount of Hemovac drainage | Postoperative 1, 2, 3 days
  CC
Total blood loss | Postoperative 1, 2, 3 days
  CC
Number of Participants with Need for transfusion | Postoperative 1, 2, 3 days
Number of Participants with Need for transfusion Deep vein thrombosis | Until postoperative 2 weeks
Visual Analog Pain Scale [0 - 10] | Preoperative & postoperative 1, 2, 3 days, 2 weeks
  Higher scores mean worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea Seoul St Mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes